CLINICAL TRIAL: NCT03507413
Title: A Prospective Randomized, Double Blind, Placebo-controlled, Safety and Efficacy Study of Metformin as add-on Therapy in Non-diabetic Patients With Abdominal Aortic Aneurysm (MetAAA Study)
Brief Title: Metformin Therapy in Non-diabetic AAA Patients
Acronym: MetAAA
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Merck Serono GmbH, Germany (Industry)
Responsible Party: Principal Investigator, Christoph Neumayer, Professor, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1479/2017
Record Dates: First submitted 2018-03-29; First posted 2018-04-25 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: abdominal aortic aneurysm; metformin; non-diabetic; placebo
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: prospective, randomized, double blind, placebo-controlled, safety and efficacy study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INVESTIGATIONAL DRUG (Active Comparator): oral metformin treatment with 2000Mg daily: Glucophage 500mg Tablet (2-0-2) daily for 1 year
  Interventions: Drug: Metformin Glucophage 500mg (IR) tablets M90
- COMPARATIVE DRUG (Placebo Comparator): Placebo matching M90 Oral Tablet treatment twice daily (2-0-2) for 1 year
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Metformin Glucophage 500mg (IR) tablets M90 — oral metformin Glucophage treatment 500 mg daily (2-0-2) for 1 year
  Other Names: Glucophage (Merck)
  Arms: INVESTIGATIONAL DRUG
Drug: Placebo Oral Tablet — Placebo Oral Tablet M90 treatment twice daily (2-0-2) for 1 year
  Other Names: Placebo (Merck)
  Arms: COMPARATIVE DRUG

SUMMARY:
A prospective randomized, double blind, placebo-controlled, safety and efficacy study of metformin as add-on therapy in abdominal aortic aneurysm (AAA)

OBJECTIVES Primary Objective

* To demonstrate treatment efficacy of metformin in AAA in comparison to placebo or active comparator, as measured by growth of the AAA maximum diameter at 12 months Secondary Objectives
* To asses inflammatory cytokines and parameters of neutrophil activation in AAA in response to metformin treatment by glucose
* insulin
* Interleukin-6
* markers of neutrophil activation (MPO, elastase, NGAL)

DETAILED DESCRIPTION:
DESIGN / PHASE Prospective, single-center, randomized, parallel group, double-blind, placebo controlled, phase IIa study STUDY PLANNED DURATION First patient First visit Year 1 1Q

Last patient First visit Year 2 4Q Last patient Last visit Year 3 2Q

CENTER(S)

* COUNTRY(IES) 1 center in 1 country Austria PATIENTS / GROUPS 170 patients in 2 groups 85 patients per group Randomization ratio 1:1 Stratification for hypertension, age, smoking habit, sex INCLUSION CRITERIA

  * Infrarenal AAA of 3.0-4.9 cm maximum diameter EXCLUSION CRITERIA
  * premenopausal female patients with a pregnancy possibility
  * patients with diabetes
  * indication for surgical AAA repair
  * life expectancy <2 years
  * contraindications for metformin, i.e. severely reduced kidney function (eGFR <30 ml/min), liver dysfunction, pancreatitis, alcohol abuse, malnutrition and decompensated heart failure STUDY PERIODS
  * 1-2 year recruitment
  * 1 year treatment
  * 12 month follow-up INVESTIGATIONAL DRUG

Metformin:

initial dose: 500 mg 1-0-1 target dose: 1000 mg 1-0-1 COMPARATIVE DRUG /CONTROL CONDITION Placebo Initial and target dose: tablets 1-0-1 CONCOMITANT MEDICATION Allowed (standard of care) EFFICACY ENDPOINTS AAA growth (in maximum diameter) over 1 year TOLERABILITY / SAFETY surgery when AAA>5.5 cm for men, > 5 cm for women

Metformin Therapy for AAA Department of Surgery, Division of Vascular Surgery Medical University of Vienna, Austria

ENDPOINTS

adverse drug reactions liver insufficiency sustained reduction of kidney function with glomeral filtration rate <30 mg/dl (upon temporary renal insufficiency, infections, exsiccosis, diarrhea and lactic acidosis, metformin treatment will only be paused)

PHARMACOKINETIC / PHARMACODYNAMIC ENDPOINTS

* glucose
* insulin
* Interleukin-6
* markers of neutrophil activation (MPO, elastase, NGAL)

QUALITY OF LIFE / PHARMACOECONOMIC ENDPOINTS gastrointestinal discomfort (as assessed in the initial drop-out phase for patient exclusion)

STATISTICAL METHODOLOGY Primary Endpoint AAA growth at 12 months in mm

Null and alternative hypotheses:

H0: Metformin does not reduce AAA growth

H1: Metformin reduces AAA growth from mean 1.7 to 0.4 mm per year Type-I and -II errors:

Significance: 5% Power: 80% 1.7±3.3 mm (mean±SD) without Metformin and 0.4±2.3 mm (mean±SD) with Metformin treatment Sample size calculation 77 per group plus 16 patients drop out Total N= 170 Statistical methodology Main analysis set: per protocol Primary endpoint: analysis of covariance adjusted for baseline AAA diameter Pharmacokinetic endpoints: analysis of covariance adjusted for baseline value. Parametric assumptions will be graphically checked with histograms.

In case of non-normal distributions analysis of covariance will be performed after a logarithmic or rank transformation.

Safety endpoints will be described by cumulative incidence curves

ELIGIBILITY:
Inclusion Criteria:

• Infrarenal AAA of 3-4.9 cm maximum diameter

Exclusion Criteria:

* premenopausal female patients with a pregnancy possibility
* patients with diabetes
* indication for surgical AAA repair
* contraindications for metformin, i.e. severly reduced kidney function (eGFR <30 ml/min), liver dysfunction, pancreatitis, alcohol abusus, malnutrition and decompensated heart failure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
AAA growth over 12 months in mm | 12 months
  AAA maximum diameter in CT scan

SECONDARY OUTCOMES:
inflammation markers IL-6 | 12 months
  inflammatory cytokines and parameters of neutrophil activation in patient plasma
glucose markers insulin and glucose | 12 months
  inflammatory cytokines and parameters of neutrophil activation in patient plasma
neutrophil markers NGAL | 12 months
  inflammatory cytokines and parameters of neutrophil activation in patient plasma
ineutrophil marker MPO | 12 months
  inflammatory cytokines and parameters of neutrophil activation in patient plasma
neutrophil marker elastase | 12 months
  inflammatory cytokines and parameters of neutrophil activation in patient plasma
AAA thrombus | 12 months
  volume of AAA thrombus

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Neumayer, MD, Principal Investigator — Medical University of Vienna; Wolf-Hans Eilenberg, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Surgery, Division of Vascular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] minimale Endnote Formatierung der Refs im Word Dokument probieren!!!
- [Derived] Klopf J, Willixhofer R, Ahmadi-Fazel D, Scheuba A, Fuchs L, Sotir A, Wanhainen A, Brostjan C, Neumayer C, Eilenberg W. MetAAA Trial Patients Receiving Metformin Therapy Show Limited Improvement in Quality of Life Compared to AAA Patients with Placebo Intake-A Double-Blind, Randomized, and Placebo-Controlled Trial. Med Sci (Basel). 2025 Nov 15;13(4):273. doi: 10.3390/medsci13040273. PMID 41283274
- [Derived] Klopf J, Willixhofer R, Scheuba A, Fuchs L, Sotir A, Wanhainen A, Brostjan C, Neumayer C, Eilenberg W. MetAAA trial patients show superior quality of life compared to patients under regular surveillance for small AAA: a single-center retrospective cohort study. Int J Surg. 2023 Apr 1;109(4):861-869. doi: 10.1097/JS9.0000000000000343. PMID 36999821